CLINICAL TRIAL: NCT00997581
Title: Apremilast Therapy for Acute Gouty Arthritis
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Colaborator withdrew support.
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AP-GOUT-PI-0038
Record Dates: First submitted 2009-10-09; First posted 2009-10-19 (Estimated); Last update posted 2018-04-02 (Actual); Status verified 2018-03

CONDITIONS: Acute Gout
Keywords: Gout
MeSH Terms: conditions — Gout | interventions — apremilast

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- apremilast (Experimental): Experimental treatment for acute gout
  Interventions: Drug: apremilast
- indomethacin (Active Comparator): Medication currently used for the treatment of acute gout
  Interventions: Drug: indomethacin SR

INTERVENTIONS:
Drug: apremilast — apremilast 20 mg taken twice daily by mouth
  Arms: apremilast
Drug: indomethacin SR — indomethacin SR 75 mg taken twice daily by mouth
  Arms: indomethacin

SUMMARY:
The purpose of the study is to learn about a possible new medicine, apremilast, for treating acute gout and compare how it works to indomethacin, a medication that has been used to treat gout for over 50 years.

In order to learn about apremilast, half the participants in this study will receive apremilast and half the participants in this study will receive indomethacin.

This study will measure the severity and duration of acute gout attacks in research participants, as well as measures of quality of life and any side effects or adverse reactions to the medication.

There will be three study visits: a screening/baseline visit on Day 1, a visit to evaluate response to treatment with study medication at Day 7, and a follow-up visit at Day 21.

DETAILED DESCRIPTION:
WITHDRAWN

ELIGIBILITY:
Inclusion Criteria:

* Must understand and voluntarily sign the informed consent
* Must have the diagnosis of gout proven by identification of urate crystals from body fluids
* Must be male age >18 years at the time of consent
* Must be able to adhere to the study visit schedule and other protocol requirements
* Must meet the following laboratory criteria:

  * Hemoglobin > 9.0 g/dL
  * White blood cell (WBC) count > 3000/μL and < 14,000/μL
  * Platelet count >100,000/μL
  * Serum creatinine < 2.0mg/dL
  * Total bilirubin < 2.0 mg/dL
  * Aspartate transaminase (AST) and alanine transaminase (ALT) <1.5 X upper limit of normal
* Males, including those who have had a vasectomy, must agree to use barrier contraception (latex condom) when engaging in sexual activity with a female of child-bearing potential (FCBP) while on study medications and for 84 days after taking the last does of the medication

Exclusion Criteria:

* Inability to provide voluntary consent
* Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he were to participate in the study or confounds the ability to interpret the data from the study
* Females
* Systemic fungal infection
* History of recurrent bacterial infection (at least 3 major infections resulting in hospitalization and/or requiring intravenous antibiotic treatment in the past 2 years
* An active infection at presentation
* Use of any investigational medication within 4 weeks prior to start of study or 5 pharmacokinetic/pharmacodynamic half-lives, whichever is longer
* Any use of corticosteroids, cyclosporine, methotrexate, cyclophosphamide, azathioprine, mycophenolate within 4 weeks prior to start of study
* Any clinically significant abnormality on 12-lead ECG screening
* Malignancy or history of malignancy (except for treated and cured basal-cell skin carcinomas > 3 years prior to screening)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-04 (Estimated); Primary Completion 2010-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Subject-reported number of swollen joints, the number of tender joints, the number of warm joints, as well as self-report pain, global assessment, and functional status. Subject-reported time to resolution of symptoms will be measured. | Day 1, Day 7 and Day 21.

SECONDARY OUTCOMES:
Safety (type, frequency, severity, and relationship of adverse events to apremilast, laboratory, ECG, physical exam or other changes) and tolerability | Day 1, Day 7 and Day 21.
Quality of Life | Assessed at Day 1, Day 7 and Day 21 study visits

CONTACTS AND LOCATIONS:
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

REFERENCES:
- [Derived] van Durme CM, Wechalekar MD, Landewe RB, Pardo Pardo J, Cyril S, van der Heijde D, Buchbinder R. Non-steroidal anti-inflammatory drugs for acute gout. Cochrane Database Syst Rev. 2021 Dec 9;12(12):CD010120. doi: 10.1002/14651858.CD010120.pub3. PMID 34882311